CLINICAL TRIAL: NCT01870271
Title: Pilotstudie Developmentally Adapted Cognitive Processing Therapy für Jugendliche Und Junge Erwachsene Mit Posttraumatischer Belastungsstörung Nach Sexualisierter Und /Oder körperlicher Gewalt (Pilot DCPT)
Brief Title: Pilot-Study DCPT for PTSD in Adolescents and Young Adults
Acronym: Pilot-DCPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Collaborators: Katholische Universität Eichstätt Ingolstadt (Unknown); Freie Universität Berlin (Other)
Responsible Party: Principal Investigator, Regina Steil, Dr., Goethe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pilot-DCPT
Record Dates: First submitted 2013-03-19; First posted 2013-06-06 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: PTSD
Keywords: PTSD; childhood sexual abuse; physical abuse; developmentally adapted cognitive processing therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DCPT (Experimental): Treatment with developmentally adapted D-CPT. 30 to 36 individual treatment sessions. Treatment sections comprise a commitment phase (5 sessions), emotion regulation phase (6 sessions), CPT (15 sessions) and a final phase targeting developmentally-related challenges (4 sessions).
  Interventions: Behavioral: Developmentally adapted cognitive processing therapy

INTERVENTIONS:
Behavioral: Developmentally adapted cognitive processing therapy

SUMMARY:
The aim of this pilot study is to evaluate the developmentally adapted cognitive processing therapy (D-CPT)in adolescents suffering from childhood abuse(CA)or physical abuse (PA) related PTSD. D-CPT's feasibility and efficacy will be examined in 20 adolescents suffering from CA or PA-related PTSD in a multicenter study (3 sites).Patients will be assessed prior to (t0), post (t1) and 6 weeks after treatment (t2). Assessments include Clinician Administered PTSD Scale (CAPS), UCLA PTSD Index (UCLA), Beck Depression Inventory (BDI), Adolescent Dissociative Experiences Scale (A-DES), and Borderline Symptom List (BSL-23).

DETAILED DESCRIPTION:
The aim of this pilot study is to evaluate the developmentally adapted cognitive processing therapy (D-CPT)in adolescents suffering from childhood sexual abuse (CA) or childhood physical abuse (PA) related PTSD. D-CPT's feasibility and efficacy will be examined in 20 adolescents suffering from CA or PA-related PTSD in a multicenter study in Berlin, Frankfurt and Ingolstadt in Germany (3 sites).Patients will be assessed prior to (t0), post (t1) and 6 weeks after treatment (t2). Assessments include Clinician Administered PTSD Scale (CAPS), UCLA PTSD Index (UCLA), Beck Depression Inventory (BDI), Adolescent Dissociative Experiences Scale (A-DES), and Borderline Symptom List (BSL-23).

ELIGIBILITY:
Inclusion Criteria:

* PTSD after CSA and/or CPA beyond the age of three (confirmed by a structured clinical interview, CAPS-CA, German Version IBS-KJ)
* PTSD must be the primary diagnosis (most severe disorder according to SCID)
* age 14 - 21 years
* living in safe conditions
* informed consent from parents/legal guardians (if under 18) and participant

Exclusion Criteria:

* current psychotic
* substance related or organic mental disorder
* acute suicidality, severe medical conditions
* mental retardation
* insufficient knowledge of German language.

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Clinician-Administered PTSD-Scale for Children and Adolescents | t0=pretreatment (baseline), t1= change from baseline at post-treatment after 20 weeks t2= change from posttreatment at 6 weeks follow-up

SECONDARY OUTCOMES:
UCLA PTSD Index (UCLA) | t0=pretreatment (baseline), t1= change from baseline at post-treatment after 20 weeks t2= change from posttreatment at 6 weeks follow-up
Beck Depression Inventory | t0=pretreatment (baseline), t1= change from baseline at post-treatment after 20 weeks t2= change from posttreatment at 6 weeks follow-up

OTHER OUTCOMES:
Borderline Symptom List (BSL-23) | t0=pretreatment (baseline), t1= change from baseline at post-treatment after 20 weeks t2= change from posttreatment at 6 weeks follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Regina Steil, PhD, Principal Investigator — Goethe University
Locations (1):
- Department of Clinical Psychology and Psychotherapy, Goethe University, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No